CLINICAL TRIAL: NCT04131348
Title: Botulinum Toxin to Avoid Component Separation in Midline Large Hernias
Acronym: BTCS01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, JOSE BUENO-LLEDÓ, Head of section, Hospital Universitario La Fe
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCS001
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Botulinum Toxin Type A; Rives Repair; Large Midline Hernia; Component Separation
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSG (Other): patients underwent open CST (component separation group or CSG)
  Interventions: Procedure: botulinum toxin type A
- BTG (Other): patients with preoperative BT administration and following open RSR (botulinum toxin group or BTG).
  Interventions: Procedure: botulinum toxin type A

INTERVENTIONS:
Procedure: botulinum toxin type A — From to December 2016 to December 2018, a single-center prospective comparative study was performed in 80 patients with LMIH at our tertiary center.

SUMMARY:
Introduction. The goal of our study was to compare results in patients with large midline incisional hernia (LMIH) using only anterior compònent separation (CST) versus preoperative botulinum toxin (BT) and following Rives repair (RSR).

Material and methods. From to December 2016 to December 2018, a prospective comparative study was performed in 80 consecutive patients with LMIH and hernia transverse diameter between 12-18 cms at our tertiary center. Two groups were prospectively analyzed: patients underwent open CST (component separation group or CSG) and patients with preoperative BT administration and following open RSR (botulinum toxin group or BTG).

DETAILED DESCRIPTION:
Multiple techniques have been described to decrease tension in the closure of the hernia defect in the large midline incisional hernias (LMIH) (1). Anterior component separation (CST) has demonstrated to accomplish primary fascial closure, while maintaining normal anatomy and physiology of the abdominal wall (2,3). However, described limitations of this technique are complications involving the skin and subcutaneous tissue, most likely caused by surgical interruption of perforating vessels during exposure of the external oblique muscle. So, CST has been related to surgical site occurrences (SSO), especially skin necrosis, up to 17% of cases, as well as recurrence rates between 7 and 18% (4).

On the other hand, botulinum toxin type A (BT) has been reported as a therapeutic option to decrease tension of a fascial closure in LMIH (5). It is a neurotoxin that causes a reversible denervation and paralisis of the lateral abdominal muscle, and has been considered as a "chemichal component separation" by some working groups (6). Our long experience about use of preoperative techniques like BT and progressive pneumperitoneum (PPP) allowed us to raise the possibility of planning the isolated use of BT in case of long transverse hernia diameters in patients with LMIH (7).

Taking advantage of the beneficial effect of the neurotoxin, we considered interesting to try to downstage the CST to other hernia repair with less morbidity, like Rives-Stoppa retromuscular repair (RSR). This technique has been traditionally considered the gold standard technique in midline hernias, especially in hernia defects with transverse diameters around or less than 10 cms, and appears to be more advantageous compared to other surgical techniques concerning complications and recurrence rates (8). RSR achieves several objectives: a tension-free closure due to extensive overlap between the prosthesis and the fascial edges, and the placement of the mesh next to the vascular-rich rectus muscles facilitates tissue incorporation and minimizing complications related to SSO (9).

The objective of our study was to compare results in two groups of patients with LMIH, using only CST versus preoperative BT plus following RSR, focusing on the SSO, possibility of primary fascial closure, length of hospital stay and hernia recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with LMIH with hernia transverse defect between 12 and 18 cms in preoperative CT scan
* grade W3 in EHS classification

Exclusion Criteria:

* patients with loss of domain hernia (Tanaka index over 20% in CT scan)
* laparoscopic approaches
* hernias not involving the midline, such as isolated flank and parastomal defects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
surgical site ocurrences after hernia repair. | two years
  focusing on the SSO (seroma, ischemia, infection) after hernia repair in both groups
primary fascial closure | two years
  possibility of free-tension closure
lenght of stay | two years
  lenght of hospital stay after hernia repair
recurrence rate | two years
  hernia recurrence rate after surgery in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Bueno-Lledo, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No